CLINICAL TRIAL: NCT04753047
Title: The Cognitive Functioning of Young Athletes (10-12 Years Old) Undertaking Various Sports Activities (Gymnastics, Football) Including Bioelectrical Brain Function
Brief Title: The Cognitive Functioning of Young Athletes Including Bioelectrical Brain Function
Status: Completed | Type: Observational
Sponsor: University of Gdansk (Other)
Responsible Party: Principal Investigator, Ilona Bidzan-Bluma, Principal Investigator, University of Gdansk
Other Study IDs: UGdansk
Record Dates: First submitted 2021-01-29; First posted 2021-02-12 (Actual); Last update posted 2022-04-20 (Actual); Status verified 2022-04

CONDITIONS: Cognitive Function
Keywords: cognitive function; sport; football; gymnastics; children

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Children practicing football: Children in late childhood (age 10-12 years) practicing sport, which is high dynamic (> 75%), and low static (<10&) and in the same time it is open skill exercise sport (football)
  Interventions: Other: No intervention
- Children practicing gymnastics: Children in late childhood (age 10-12 years) practicing sport, which is low dynamic (<50%), high static (>30%) and in the same time it is closed skill exercise sport (sport gymnastics)
  Interventions: Other: No intervention
- Comparative group: A comparative group of children that do not attend sport classes or sports clubs, but carrying out sports activity and / or in other areas
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
The project focuses on two central issues:

1. The impact of intensity of sport on the cognitive functioning and brain waves of children in late childhood (10-12 years old);
2. The specific impact of individual forms of sporting competitions classified according to dynamic, static components as well as closed / open skill exercise. The variables will be age, gender, and fluid intelligence. Additionally, children's temperament will be examined in order to assess its relationship with the preferences for choosing a particular type of sport activity and the intensity of this activity.

ELIGIBILITY:
Inclusion Criteria:

- Polish-speaking children

Exclusion Criteria:

* mental illness;
* non-Polish speaking children

Ages: 10 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Gender Based: Yes
Study Population: The participants will be recruited for research via Szkoły Mistrzostwa Sportowego [Sports Championship Schools] (criterion groups), sports clubs, as well as by establishing contact with other primary schools. Selecting 40 - 45 people aged 10-12 for each of the 2 control groups differentiated by the dynamic, static factor and nature of the sport close / open skill and for the comparative group of 40-45 children who are cognitively stimulated through physical activity and / or otherwise.
  They will be enrolled to the study after giving their and their parents written consent to participate in the study.
Sampling Method: Non-Probability Sample
Enrollment: 179 (Actual)
Dates: Start 2020-01-02 (Actual); Primary Completion 2022-01-02 (Actual); Study Completion 2022-01-02 (Actual)

PRIMARY OUTCOMES:
Attention | Baseline
  - PU1 Battery (Borkowska, SajewiczRadtke, Lipowska, Kalka, 2016) - attention (the ability to orientate on stimulus, motor speed, maintain attention on the visual stimulus, distinguishing significant and non-significant material). Higher score means better attention.
Brain Waves | Baseline
  - EEG Biofeedback - bioelectric recording of brain activity from a centrally placed electrode to measure fast brainwaves (Alpha, Beta1, Beta2) and slow brainwaves (Delta, Theta)
Short-term memory of verbal material material | Baseline
  - PU1 Battery (Borkowska, SajewiczRadtke, Lipowska, Kalka, 2016). Higher score means better short-term memory of verbal material
Visual-spatial material | Baseline
  - PU1 Battery (Borkowska, SajewiczRadtke, Lipowska, Kalka, 2016). Higher score means better visual-spatial material.
Executive functions | Baseline
  - PU1 Battery (Borkowska, SajewiczRadtke, Lipowska, Kalka, 2016). Higher score means better executive functions.
Language functions | Baseline
  - PU1 Battery (Borkowska, SajewiczRadtke, Lipowska, Kalka, 2016). Higher score means better language functions.
Episodic memory of visual-spatial material | Baseline
  - Diagnosis of Brain Injury (DUM) (Weidlich, Lamberti, 1996) [assessment of episodic memory of visual-spatial material (the rate of acquiring new information, the process of consolidation - the ability to transfer information from short-term to long-term memory)]. Higher score means better episodic memory of visual-spatial material (maximal points: 54, minimal: 0).

SECONDARY OUTCOMES:
Sports Intensity by International Physical Activity Questionnaire (in a modified version, relating to children) (Biernat, 2007) | Baseline
  Higher scores mean a better physical activity. In test there are 3 categories of activity: insufficient (less than 600), sufficient (600 - 1500 or 600 - 3000) or high (more than 1500 or 3000 MET-min / week)
Intelligence by CFT 20-R, The Culture Fair Intelligence Test (CFIT) - version 2, part 1 only (Cattell, Weiss, adapt. Stańczak,2013) | Baseline
  Measurement of fluid intelligence. Higher score means higher fluid intelligence (maximum number of points: 56, minimal: 0).
Temperament by EAS Buss & Plomin Questionnaire (Buss, Plomin, 1997) | Baseline
  A questionnaire for parents, coaches, teachers. It consists of 20 items - statements, which suitableness is rated by the subject on a five-point scale (from "Never true" to "Always true"). This version has four scales: Shyness, Sociability, Activity, and Emotionality and has 20 items relating to each of the 4 temperaments. There is a 5-point rating scale (from 1: "not characteristic or typical of your child" to 5 : "very characteristic or typical of your child"). These scores belong to each temperament and they are summed.

CONTACTS AND LOCATIONS:
Overall Officials: Ilona Bidzan-Bluma, MS, Principal Investigator — University of Gdansk
Locations (2):
- Poland (2):
  - University of Gdansk, Gdansk, Gdansk
  - University of Gdansk, Gdansk

REFERENCES:
- [Derived] Bidzan-Bluma I. Twin-To-Twin Transfusion Syndrome Donor and Recipient and Their Subsequent Cognitive Functioning in Late Childhood as Juvenile Athletes-A Case Study. Int J Environ Res Public Health. 2021 Mar 4;18(5):2545. doi: 10.3390/ijerph18052545. PMID 33806653